CLINICAL TRIAL: NCT03747848
Title: A Treatment Protocol for Management of Fatigue in Parkinson's Disease Using Cognitive Behavioral Therapy
Brief Title: Treatment Protocol for PD Fatigue Management With CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1401
Record Dates: First submitted 2018-10-31; First posted 2018-11-20 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: fatigue; cognitive behavioral therapy
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT group (Experimental): Subjects will participate in group treatment sessions (once a week for six weeks).
  Interventions: Behavioral: CBT group

INTERVENTIONS:
Behavioral: CBT group — Each interested individual will complete eligibility screening, consent form, and pre-intervention assessment. Demographic information such as gender, age, and number of years since diagnosis of PD will be collected. This investigator will implement the treatment program by meeting with the participants in groups, once a week, for six weeks. Group meetings will encourage interaction and support among group participants. Program content includes encouraging physical exercise with higher intensity, changing poor sleeping hygiene habits, stress management, and encouraging utilization of social support.

SUMMARY:
Fatigue affects more than half of people living with Parkinson's disease. Despite its prevalence, treatment options remain limited. To improve patient outcome, a group treatment protocol was developed for PD fatigue management primarily using cognitive behavioral therapy. The program focuses on assisting individuals with PD who experience fatigue to establish proper sleep hygiene habits and a physical exercise routine to meet the end goal of reducing fatigue. The aim of the group is to change negative thoughts and behavior regarding changing sleep hygiene habits and exercise behavior into positive ones. This is a feasibility project that aims to explore the feasibility of this protocol as well as to produce a treatment protocol that is able to be replicated by other occupational therapists and health professionals who serve the PD population.

DETAILED DESCRIPTION:
PD is the second most common neurodegenerative disorder in the United States. Although PD is typically classified as a movement disorder, the non-motor symptoms (NMS) also have a negative impact on quality of life. Among the NMS, fatigue is one of the most reported and bothersome symptoms, even at the early stage of the disease. Currently there are not any clear pharmacological or rehabilitative recommendations for managing PD related fatigue.

The purpose of this study is to evaluate the feasibility and effectiveness of a developed treatment protocol specifically adapted to the Parkinson's population to address fatigue symptoms based on the best available evidence. This is a one-group, pre-post, feasibility study. It is hypothesized that an establishment of a proper sleep hygiene routine and a moderate- to intensive-exercise routine three times a week will decrease Parkinson's disease (PD) related fatigue and improve health-related quality of life. The treatment protocol focuses on assisting individuals with PD experiencing fatigue to improve sleep hygiene habits and establish physical exercise routine using cognitive behavioral therapy in a group format. Through this study, the designed program will be evaluated to determine if it will decrease self-perceived fatigue level and to improve health-related quality of life among community dwelling people with PD.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must be diagnosed with PD, without the diagnosis of Lewy Body dementia. Atypical parkinsonism such as Progressive Supranuclear Palsy, Corticobasal Degeneration, and Multiple System Atrophy are excluded.
2. All participants of the program are community dwelling.
3. Subjects must age between 21 and 80. There is no gender limitation.
4. All subjects report feeling sense of fatigue.
5. Because the intervention involves encouraging individuals to participate in highly-intense physical exercise or multimodal moderately-intense physical exercise, cardiovascular clearance from each participant's physician (either primary care, internist, or cardiologist) is required. See attachment for cardiovascular clearance letter.
6. Because cognitive behavioral therapy will be used in the interventions, and safety judgment is required when choosing an appropriate physical exercise during interventions, participants must present with adequate cognitive capacity. The Montreal Cognitive Assessment (MoCA) will be used to determine if the individual meets the cognitive criteria. MoCA score must be 24 or above, or 21 to 23 with an accompany of a caregiver to participate (MoCA total score is 30). In PD, individuals with mild neurocognitive disorder (NCD), with MoCA score 21 to 23, are able to perform everyday activities independently, although with greater effort, compensatory strategies, or accommodation

Exclusion Criteria:

1. MoCA score 22 or below
2. Unable to obtain physician clearance for exercise participation
3. Diagnosis of Lewy Body dementia. Atypical parkinsonism

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | 0-week, 6-week, 12-week. This is to measure the change between three points. 0-week indicates pre-treatment status; 6-week indicates post-treatment status immediately; and 12-week indicates long-term status
  Measurement of self-report fatigue level. There are 21 items on a 5-point scale- subjects rate from "Never"=0, "Rarely"=1, "Sometimes"=2, "Often"=3, to "Always"=4.
  MFIS can be aggregated into three subscales: physical, cognitive, and psychosocial.
  Total scores range from 0 to 84 (physical subscale: 0-36, cognitive subscale: 0-40, psychosocial subscale 0-8), with a higher score representing a greater impact of fatigue on a person's activities.)

SECONDARY OUTCOMES:
Sleep Hygiene Index (SHI) | 0-week, 6-week, 12-week. This is to measure the change between three points. 0-week indicates pre-treatment status; 6-week indicates post-treatment status immediately; and 12-week indicates long-term status
  Measurement of self-report sleep hygiene behavior. There are 13-item, on a five-point scale ranging from "never"=0, "rarely"=1, "sometimes"=2, "frequent"=3, to "always"=4.
  Total scores range from 0 to 52, with a higher score representing poorer sleep hygiene.
Parkinson's Sleep Scale (PDSS-2) | 0-week, 6-week, 12-week. This is to measure the change between three points. 0-week indicates pre-treatment status; 6-week indicates post-treatment status immediately; and 12-week indicates long-term status
  Measurement of self-report quality of sleep. There are 15 items about various sleep and nocturnal disturbance; rated on a 5-point scale ranging from "never"=0, occasional"=1, "sometimes"=2, "often"=3 to "very often"=4.
  Total scores range from 0 to 60, with a higher score representing poorer sleep quality.
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 0-week, 6-week, 12-week. This is to measure the change between three points. 0-week indicates pre-treatment status; 6-week indicates post-treatment status immediately; and 12-week indicates long-term status.
  Measurement of self-report health-related quality of life. There are 39 items, grouped in 8 subscales: Mobility (10 items), Activities of daily living (6 items), Emotional well-being (6 items), Stigma (4 items), Social support (3 items), Cognitions (4 items), Communication (3 items), Bodily discomfort (3 items). Total score is calculated for outcome.
  Subjects rated on a 5-point scale, ranging from "Never"=0, "occasionally"=1, "sometimes"=2, "often"=3 to "always"=4. Each dimension total scores range from 0-100, with a higher score representing worse quality of life.
  Dimension score is sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Wan-Albert, MS, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States